CLINICAL TRIAL: NCT04843007
Title: Alvopem® (Pemetrexed) Safety Assessment in Patients With Non-small Cell Lung Cancer and Malignant Pleural Mesothelioma
Brief Title: Alvopem® (Pemetrexed) Safety Assessment
Status: Completed | Type: Observational
Sponsor: NanoAlvand (Industry)
Responsible Party: Sponsor
Other Study IDs: ALVOPEM.NA.AK.95 (IV)
Record Dates: First submitted 2021-04-07; First posted 2021-04-13 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-08

CONDITIONS: Non Small Cell Lung Cancer; Malignant Pleural Mesothelioma
Keywords: NSCLC; Observational study; pemetrexed; PMS; Safety
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Mesothelioma, Malignant | interventions — Pemetrexed

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NanoAlvand Pemetrexed: 500 mg/m^2 pemetrexed, intravenous (IV) infusion
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed — Alvopem® was administered every 3 weeks with a dose of 500 mg/m^2
  Other Names: Alvopem®

SUMMARY:
The present study was a phase IV, post-marketing, observational study for safety evaluation of Alvopem® use in Iranian patients with non-small cell lung cancer and malignant pleural mesothelioma. No control groups were included in the study design.

The primary objective of this study was safety assessment, including the incidence of adverse events (AEs).

DETAILED DESCRIPTION:
The present study was a phase IV, post-marketing, observational study for safety evaluation of Alvopem® use in Iranian patients with non-small cell lung cancer and malignant pleural mesothelioma.

Data was gathered in one booklet, which had 6 different periods. The patients' information assessed after each injection, every 3 weeks. These booklets were completed by designated physicians.

The primary objective of this study was safety assessment, including the incidence and intensity of AEs and serious adverse events (SAEs).

This study was single arm and the sample size of this study was 199 patients.

ELIGIBILITY:
Inclusion Criteria: Patients diagnosed with non-small cell lung cancer and malignant pleural mesothelioma under chemotherapy regimens with Alvopem® were enrolled in the study.

Exclusion Criteria: There were no exclusion criteria for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with non-small cell lung cancer and malignant pleural mesothelioma were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Khosravi, Assoc. Prof., Principal Investigator — National Research Institute of Tuberculosis and Lung Disease (NRITLD)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Seifi S, Salimi B, Monfared ZE, Sabahi C, Kafi H, Khosravi A. Alvopem(R) (pemetrexed) safety assessment in patients with non-small cell lung cancer or malignant pleural mesothelioma: a post-marketing surveillance. J Pharm Policy Pract. 2023 Jan 25;16(1):16. doi: 10.1186/s40545-023-00524-5. PMID 36698207

RESULTS

PARTICIPANT FLOW:
Groups:
- NanoAlvand Pemetrexed: 500 mg/m^2 pemetrexed, IV infusion
  Pemetrexed: Alvopem® was administered every 3 weeks with a dose of 500 mg/m^2
Period: Overall Study
Arm/Group | NanoAlvand Pemetrexed
Started | 199
Completed | 198
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | NanoAlvand Pemetrexed
Number analyzed (Participants) | 198
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.11 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 130
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 198
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: Kg] | 66.93 (14.74)
Height [Mean (Standard Deviation); unit: cm] | 166.44 (9.88)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] | 1.75 (0.21)
Smokers [Count of Participants; unit: Participants] | 132
Diagnosis [Count of Participants; unit: Participants]
  NSCLC | 186
  MPM | 12
Serum Creatinine (SCr) [Mean (Standard Deviation); unit: mg/dL] | 1.02 (0.22)
Bilirubin [Mean (Standard Deviation); unit: mg/dL] | 0.46 (0.30)
Blood Urea Nitrogen (BUN) [Mean (Standard Deviation); unit: mg/dL] | 31.24 (10.34)
Aspartate Aminotransferase (AST) [Mean (Standard Deviation); unit: units/L] | 23.78 (21.72)
Alanine Aminotransferase (ALT) [Mean (Standard Deviation); unit: units/L] | 23.99 (17.83)
Platelet (PLT) [Mean (Standard Deviation); unit: cells/μL] | 324653 (109183)
White Blood Cell (WBC) [Mean (Standard Deviation); unit: cells/μL] | 10519 (4920)
Neutrophil [Mean (Standard Deviation); unit: cells/μL] | 7743 (4541)
Hemoglobin (Hb) [Mean (Standard Deviation); unit: g/dL] | 12.68 (1.90)

OUTCOME MEASURES:

1. Primary Outcome: Safety Assessment Including Treatment-related Adverse Events (Number of Participants Who Experienced at Least One Adverse Event (AE) or One Serious Adverse Event (SAE))
Description: In this study, number of participants who experienced at least one adverse event (AE) or one serious adverse event (SAE) were assessed. The intensity of AEs was graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 and terminology for AEs was chosen according to the Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term. Also, intensity, seriousness, onset of AEs, and interventions for management of the adverse events were documented in the booklet. For each AE, data was summarized using system organ class and preferred term of AEs and SAEs. Moreover, causality assessment was done based on the World health organization-Uppsala Monitoring Centre (WHO-UMC) system.
Time Frame: This outcome was assessed throughout the study, up to 18 weeks (6 chemotherapy cycles). The duration of treatment was at the physicians' discretion based on the patient's condition
Population: The safety population is defined as all patients who received at least one dose of the study drug. In this study, a total of 199 patients with non-squamous non-Small cell lung cancer (NSCLC) or malignant pleural mesothelioma (MPM) were enrolled. However, one patient was excluded from the safety analysis due to the absence of a recorded diagnosis, resulting in a safety population of 198 individuals.
Measure: Count of Participants; unit: Participants
Arm/Group | NanoAlvand Pemetrexed
Number analyzed (Participants) | 198
Participants | 190

ADVERSE EVENTS:
Time Frame: Three years and half
Arm/Group | NanoAlvand Pemetrexed
All-Cause Mortality (participants affected / at risk) | 28/198
Serious Adverse Events (participants affected / at risk) | 50/198
Other Adverse Events (participants affected / at risk) | 190/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NanoAlvand Pemetrexed (N=198)
Anaemia (Blood and lymphatic system disorders) | 50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NanoAlvand Pemetrexed (N=198)
Anaemia (Blood and lymphatic system disorders) | 177
leukopenia (Blood and lymphatic system disorders) | 49
neutropenia (Blood and lymphatic system disorders) | 57
Thrombocytopenia (Blood and lymphatic system disorders) | 20
Alanine aminotransferase increased (Investigations) | 20
Aspartate aminotransferase increased (Investigations) | 12
Creatinine renal clearance decreased (Investigations) | 48
Renal disorder (Renal and urinary disorders) | 1
Drug intolerance (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT04843007/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT04843007/SAP_001.pdf